CLINICAL TRIAL: NCT01827670
Title: A Clinical Study Investigating the Efficacy of a Dentifrice in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: Investigating the Efficacy of a Dentifrice in Providing Long Term Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01685
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.454% stannous fluoride dentifrice (Experimental): Participants to brush whole mouth with 1-inch strip of the test dentifrice (0.454% SnF) for one timed minute, followed by rinsing with 5 milliliter (mL) of water.
  Interventions: Drug: Stannous fluoride
- 0.76% sodium monofluorophosphate dentifrice (Active Comparator): Participants to brush whole mouth with 1-inch strip of the control dentifrice (0.76% NaMFP) for one timed minute, followed by rinsing with 5 mL of water.
  Interventions: Drug: Sodium monofluorophosphate

INTERVENTIONS:
Drug: Stannous fluoride — Test dentifrice containing 0.454% SnF
  Arms: 0.454% stannous fluoride dentifrice
Drug: Sodium monofluorophosphate — Control dentifrice containing 0.76% w/w Sodium Monofluorophosphate [1000 parts per million (ppm) fluoride]
  Arms: 0.76% sodium monofluorophosphate dentifrice

SUMMARY:
Clinical studies have demonstrated long term relief from dentine hypersensitivity with twice daily brushing of a toothpaste containing stannous fluoride in comparison to marketed (negative) controls. The aim of this study is to evaluate the effectiveness of a stannous fluoride dentifrice in the treatment of dentinal hypersensitivity compared to a marketed (negative) control, over a period of 56 days (8 weeks) with twice daily brushing.

ELIGIBILITY:
Inclusion Criteria:

* Participants with self-reported history of dentinal hypersensitivity lasting more than 6 months but not more than 10 years.
* Participants with minimum of 20 natural teeth.
* At screening, a minimum of two accessible teeth (incisors, canines, premolars) that meet all of the following criteria.

  1. Teeth showing signs of facial/cervical gingival recession and/or signs of erosion or abrasion.
  2. Teeth with Gingival Index score ≤1 and a clinical mobility of ≤1.
  3. Teeth that are determined to be sensitive by the subject following a 1 second air blast to the cervical margin.

Exclusion Criteria:

* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes dry mouth.
* Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening.
* Participant using of a desensitising dentifrice within 6 weeks of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

REFERENCES:
- [Derived] Parkinson CR, Jeffery P, Milleman JL, Milleman KR, Mason S. Confirmation of efficacy in providing relief from the pain of dentin hypersensitivity of an anhydrous dentifrice containing 0.454% with or without stannous fluoride in an 8-week randomized clinical trial. Am J Dent. 2015 Aug;28(4):190-6. PMID 26437498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Participants with a minimum of two non-adjacent sensitive teeth (incisors, canines or pre-molars) with a Schiff Sensitivity Score(following an air blast stimulus) of ≥ 2 and a tactile threshold (Yeaple probe) of ≤ 20 grams (g) force were enrolled in this study.
Groups:
- Control Dentifrice (0.76% Sodium Monofluorophosphate): Participants dosed the toothbrush with at least a 1-inch strip of the control dentifrice [0.76% weight for weight (w/w) Sodium Monofluorophosphate] and brushed whole mouth for one timed minute. Participants were permitted to rinse after each brushing with 5 milliliter (mL) potable water (kept at room temperature) for a maximum 5 timed seconds .
- Test Dentifrice (0.454% Stannous Fluoride): Participants dosed the toothbrush with at least a 1-inch strip of the test dentifrice (0.454 % w/w Stannous Fluoride) and brushed whole mouth for one timed minute, ensuring they brushed all sensitive areas of their teeth. Participants were permitted to rinse after each brushing with 5 mL potable water (kept at room temperature) for a maximum 5 timed seconds
Period: Overall Study
Arm/Group | Control Dentifrice (0.76% Sodium Monofluorophosphate) | Test Dentifrice (0.454% Stannous Fluoride)
Started | 60 | 59
Completed | 57 | 56
Not Completed | 3 | 3
Not completed — Withdrawal of Consent | 3 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Dentifrice (0.76% Sodium Monofluorophosphate): Participants dosed the toothbrush with at least a 1-inch strip of the control dentifrice [0.76% weight for weight (w/w) Sodium Monofluorophosphate] and brushed whole mouth for one timed minute. Participants were permitted to rinse after each brushing with 5 milliliter (mL) potable water (kept at room temperature) for a maximum 5 timed seconds.
- Total: Total of all reporting groups
Arm/Group | Control Dentifrice (0.76% Sodium Monofluorophosphate) | Test Dentifrice (0.454% Stannous Fluoride) | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (12.27) | 42.2 (11.27) | 42.6 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 (75.4) | 46 (80.7) | 89
  Male | 14 (24.6) | 11 (19.3) | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Schiff Sensitivity Score
Description: The examiner conducted the evaporative air sensitivity assessment and scored the subject's response to the sensitivity stimulus using the four-point categorical Schiff Sensitivity Scale (SSS).
  Score 0 = Subject does not respond to air stimulus Score 1 = Subject responds to air stimulus, but does not request discontinuation of stimulus Score 2 = Subject responds to air stimulus, and requests discontinuation or moves from stimulus Score 3 = Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation
Time Frame: Baseline-Week 8
Population: Efficacy assessments were based on intent-to-treat (ITT) population, defined as all randomized participants, administered at least one dose of study treatment providing at least one post-baseline assessment of efficacy. One participant was lost to follow-up after visit 2 in test dentifrice group but was included in the efficacy analysis at visit 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Control Dentrifice (0.76% Sodium Monofluorophosphate): Participants dosed the toothbrush with at least a 1-inch strip of the control dentifrice [0.76% weight for weight (w/w) Sodium Monofluorophosphate] and brushed whole mouth for one timed minute. Participants were permitted to rinse after each brushing with 5 milliliter (mL) potable water (kept at room temperature) for a maximum 5 timed seconds.
- Test Dentrifice (0.454% Stannous Fluoride): Participants dosed the toothbrush with at least a 1-inch strip of the test dentifrice (0.454 % w/w Stannous Fluoride) and brushed whole mouth for one timed minute, ensuring they brushed all sensitive areas of their teeth. Participants were permitted to rinse after each brushing with 5 mL potable water (kept at room temperature) for a maximum 5 timed seconds.
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride)
Number analyzed (Participants) | 57 | 57
Score on a scale
  Schiff Sensitivity Score at Baseline | 2.26 (0.379) | 2.25 (0.355)
  Schiff Sensitivity Score at Week 8 | 2.09 (0.628) | 0.78 (0.687)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride); The principal null hypothesis tested was as follows: H0: The change from baseline was same for both treatments. H1: The change from baseline was different for both the treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model: Treatment as fixed factor & baseline Schiff score as covariate; Adjusted Mean = -1.29, 95% CI 2-sided [-1.53 to -1.06] — Difference was 0.454% stannous fluoride minus 0.76% sodium monofluorophosphate such that a negative difference favours first named treatment

2. Secondary Outcome: Mean Change From Baseline in Schiff Sensitivity Score
Description: as for outcome 1
Time Frame: Baseline-Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride)
Number analyzed (Participants) | 57 | 57
Score on a Scale
  Schiff Sensitivity Score at Baseline | 2.26 (0.379) | 2.25 (0.355)
  Schiff Sensitivity Score at Week 4 | 2.10 (0.601) | 1.27 (0.598)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model: Treatment as fixed factor & baseline Schiff score as covariate; Adjusted Mean = -0.81, 95% CI 2-sided [-1.00 to -0.62] — Difference was 0.454% Stannous Fluoride minus 0.76% Sodium MonoFluorophosphate such that a negative difference favored first named treatment

3. Secondary Outcome: Mean Change From Baseline in Tactile Sensitivity
Description: The examiner assessed the tactile sensitivity of eligible teeth using a Yeaple probe. The constant pressure applied by Yeaple probe probe allowed the examiner to vary the force applied to the dentin surface from 10g to an upper threshold of 80g, in increments of 10g. The greater the pressure the participant was able to tolerate, the less sensitive the tooth was considered. Testing began at 10g and increased by 10g, with each successive challenge, until either a "yes" response (pain was elicited) was recorded or the maximum force has been reached.
Time Frame: Baseline-Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride)
Number analyzed (Participants) | 57 | 57
Grams
  Tactile Threshold at Baseline (g) | 10.1 (0.66) | 10.4 (1.43)
  Tactile Threshold at Week 8 (g) | 14.6 (13.77) | 41.6 (25.85)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model: Treatment and baseline Schiff stratification value as fixed factor and baseline tactile threshold as covariate; Adjusted Mean Difference = 27.2, 95% CI 2-sided [19.4 to 35.1] — Difference was 0.454% Stannous Fluoride minus 0.76% Sodium MonoFluorophosphate such that a positive difference favours first named treatment

4. Secondary Outcome: Mean Change From Baseline in Tactile Sensitivity
Description: as for outcome 3
Time Frame: Baseline-Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Groups:
- Control Dentrifice (0.76% Sodium Monofluorophosphate): Participants dosed the toothbrush with at least a 1-inch strip of the control dentifrice [0.76% weight for weight (w/w) Sodium Monofluorophosphate] and brushed whole mouth for one timed minute. Participants were permitted to rinse after each brushing with 5 mililiter (mL) potable water (kept at room temperature) for a maximum 5 timed seconds
- Test Dentrifice (0.454% Stannous Fluoride Dentifrice): Participants dosed the toothbrush with at least a 1-inch strip of the test dentifrice (0.454% w/w Stannous Fluoride) and brushed whole mouth for one timed minute, ensuring they brushed all sensitive areas of their teeth. Participants were permitted to rinse after each brushing with 5 mL potable water (kept at room temperature) for a maximum 5 timed seconds
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride Dentifrice)
Number analyzed (Participants) | 57 | 57
Grams
  Tactile Thresold (g) at Baseline | 10.1 (0.66) | 10.4 (1.43)
  Tactile Thresold (g) at Week 4 | 15.8 (14.78) | 24.6 (17.53)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride Dentifrice); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0138, ANCOVA; [statistical method as in outcome 3, analysis 1]; Adjusted Mean = 7.5, 95% CI 2-sided [1.6 to 13.4] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Mean Change in Dentinal Hypersensitivity After 4 Weeks as Measured by Visual Analog Scale (VAS)
Description: The subject rated the intensity of their response to the evaporative air stimulus by rating the intensity of their response to the stimulus using a 100 millimeter (mm )VAS Scale 0 is No Pain and 100 is Worst Pain Imaginable A trained member of staff measured the line segment marked off in mm and recorded this measurement in the CRF
Time Frame: Baseline-Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Test Dentrifice (0.454% Stannous Fluoride): Participants dosed the toothbrush with at least a 1-inch strip of the test dentifrice (0.454% w/w Stannous Fluoride) and brushed whole mouth for one timed minute, ensuring they brushed all sensitive areas of their teeth. Participants were permitted to rinse after each brushing with 5 mL potable water (kept at room temperature) for a maximum 5 timed seconds.
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride)
Number analyzed (Participants) | 57 | 57
Score on a Scale
  VAS Score at Baseline | 58.40 (21.661) | 58.26 (21.099)
  VAS Score at week 4 | 50.32 (23.257) | 38.09 (21.612)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA; From ANCOVA model: Treatment and baseline Schiff stratification value as fixed factor and baseline VAS as covariate; Adjusted Mean = -12.14, 95% CI 2-sided [-18.51 to -5.77] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Mean Change in Dentinal Hypersensitivity After 8 Weeks as Measured by Visual Analog Scale (VAS)
Description: as for outcome 5
Time Frame: Baseline - Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Control Dentrifice (0.76% Sodium Monofluorophosphate) | Test Dentrifice (0.454% Stannous Fluoride)
Number analyzed (Participants) | 57 | 57
Score on a Scale
  VAS Score at Baseline | 58.40 (21.661) | 58.26 (21.099)
  VAS Score at Week 8 | 43.94 (23.996) | 22.17 (22.299)
Statistical Analysis 1: Comparison: Control Dentrifice (0.76% Sodium Monofluorophosphate) vs Test Dentrifice (0.454% Stannous Fluoride); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model: Treatment and baseline Schiff stratification value as fixed factor and baseline VAS as covariate; Adjusted Mean = -21.82, 95% CI 2-sided [-29.55 to -14.09] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All Adverse events encountered or spontaneously reported following use of dentifices were reported at Baseline visit(Visit 2), 28 days(Visit 3) and Visit 4(Day 56)
Arm/Group | Control Dentifrice (0.76% Sodium Monofluorophosphate) | Test Dentifrice (0.454% Stannous Fluoride)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 2/60 | 1/59
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Dentifrice (0.76% Sodium Monofluorophosphate) (N=60) | Test Dentifrice (0.454% Stannous Fluoride) (N=59)
Dysgeusia (General disorders) | 0 (0) | 1 (1)
Mouth Injury (General disorders) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.